CLINICAL TRIAL: NCT04970459
Title: Constitution of a Biological Collection to Study the Pathophysiology in Marfan Syndrome and Related Syndromes and to Identify Predictive Factors of Disease Progression
Brief Title: Biological Collection for Marfan and Related Syndromes
Acronym: MARFANS
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Other Study IDs: RC31/21/0178
Record Dates: First submitted 2021-07-09; First posted 2021-07-21 (Actual); Last update posted 2024-03-29 (Actual); Status verified 2024-03

CONDITIONS: Marfan Syndrome
Keywords: Biological collection; Marfan syndrome; Marfan associated syndromes
MeSH Terms: conditions — Marfan Syndrome | interventions — Urination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — extra sample of blood and urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with Marfan syndrome or related syndromes: Children aged at least 3 years old or adult with Marfan syndrome or related syndromes
  Interventions: Biological: collection of samples of blood and urine

INTERVENTIONS:
Biological: collection of samples of blood and urine — extra samples of blood and urine will be collected and stored for research utilisation

SUMMARY:
The present study will establish a collection of biological samples from Marfan patients or with associated diseases to be used for research purposes only, with due respect for confidentiality.

DETAILED DESCRIPTION:
Marfan syndrome is an autosomal dominant disease (incidence 1/5000) characterized by ocular, cardiac and skeletal abnormalities. More recently, a decrease in fat and muscle mass has been demonstrated, associated with a decrease in exercise endurance, causing a significant deterioration in the quality of life. Little is known about the pathophysiology of these symptoms. Patients with Marfan syndrome or related diseases are followed at the children's hospital as part of the Rare Diseases Reference Centre (CRMR) for Marfan syndrome at the Toulouse University Hospital. During regular check-up visits, an extra sample of blood and urine will be collected and stored for research utilisation with the patient's consent. The ultimate objective of this collection is to provide available biological resources to facilitate the development of subsequent studies aimed at better characterizing the multisystemic disorders in Marfan syndrome, to understand the pathophysiology of the disease, and to identify biological factors that predict the severity and progression of the disease. The possibility of having systematically collected biological resources will make it possible to answer certain questions more quickly depending on the progress of research.

ELIGIBILITY:
Inclusion Criteria:

* Children aged at least 3 years old or adult with Marfan syndrome or related syndromes
* Patients affiliated to or beneficiaries of a social security scheme
* Patients able to receive information on the progress of the study and understand the information form to participate in the study. That implies to master the French language and not to be subject to a restriction of rights by the judicial authorities
* Patients or legal representative who have given their consent to participate in the study (expression of no objection)

Exclusion Criteria:

* Patients subject to a legal protection measure (guardianship, curators, or safeguard of justice)
* Pregnant or breastfeeding women

Ages: 3 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients followed at the Rare Diseases Reference Centre (CRMR) for Marfan syndrome at the Toulouse University Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2022-01-24 (Actual); Primary Completion 2026-08-07 (Estimated); Study Completion 2031-08-07 (Estimated)

PRIMARY OUTCOMES:
Constitution of a biological collection from patients with Marfan or related syndromes. | Day 0
  extra sample of blood and urine will be collected
Constitution of a biological collection from patients with Marfan or related syndromes. Collection of samples at inclusion. | during the intervention/procedure/surgery
  extra sample of blood and urine will be collected

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Edouard, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- Purpan University Hospital, Toulouse, France

IPD SHARING:
Plan to Share IPD: No